CLINICAL TRIAL: NCT01303406
Title: A Phase IIIb Double-Blind, Randomised, Placebo-Controlled Study of Patient Reported Outcomes in Friedreich's Ataxia Patients After Withdrawal From Treatment With Idebenone
Brief Title: Patient Reported Outcomes in Friedreich's Ataxia Patients After Withdrawal From Treatment With Idebenone (PROTI)
Acronym: PROTI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNT-III-004
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Friedreich's Ataxia
Keywords: randomized withdrawal; idebenone; friedreich's ataxia; Miconos; Patient reported outcome; ICARS
MeSH Terms: conditions — Friedreich Ataxia | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Following the body weight, patients will be allocated to one of the following regimen:
  Placebo Patients < 45 kg - 3 tablets 3 times a day with meals
  Placebo Patients > 45 kg - 5 tablets 3 times a day with meals
  Interventions: Drug: Placebo
- idebenone (Experimental): Following the body weight, patients will be allocated to one of the following regimen:
  Idebenone Patients < 45 kg - 3 tablets 3 times a day with meals
  Idebenone Patients > 45 kg - 5 tablets 3 times a day with meals
  Interventions: Drug: Idebenone

INTERVENTIONS:
Drug: Idebenone — All PROTI patients randomised to idebenone treatment will receive high dose idebenone. This is defined according to body weight. In patients weighing 45 kg or less, it is 1350 mg/day (3 x 150 mg tablets three times per day with meals). In patients weighing more than 45 kg, it is 2250 mg/day (5 x 150 mg tablets three times per day with meals).
  Other Names: Catena (approved name in Canada)
  Arms: idebenone
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase IIIb Double-Blind, Randomised, Placebo-Controlled Study. The aim is to further investigate the effects of idebenone in patients with Friedreich's ataxia.

The objective of the PROTI study is to establish whether patients can correctly determine which treatment assignment (placebo or idebenone) they received during the randomised phase of the trial, and identify any potential changes on symptoms or activities.

ELIGIBILITY:
Inclusion Criteria:

* Completion of V5 (Month 12), V6 (Month 18), or V7 (Month 24) in the MICONOS extension study
* Patients who in the opinion of the investigator are able to comply with the requirements of the study
* Body weight ≥ 25kg
* Negative urine pregnancy test

Exclusion Criteria:

* AE during the course of the MICONOS extension study which in the opinion of the investigator is attributable to idebenone and precludes further treatment with idebenone
* Clinically significant abnormalities of clinical haematology or biochemistry including, but not limited to, elevations greater than 1.5 times the upper limit of normal SGOT, SGPT or creatinine
* Parallel participation in another clinical drug trial
* Pregnancy or breast-feeding
* Abuse of drugs or alcohol
* Any change of concomitant medication within the last 30 days that in the opinion of the investigator the intake could negatively impact the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Giunti, M.D, Principal Investigator — Institute of Neurology, The National Hospital, University College London
Locations (6):
- Innsbruck, Austria
- Germany (3):
  - Bonn
  - München
  - Tübingen
- Groningen, Netherlands
- The National Hospital, University College London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Following the body weight, patients will be allocated to one of the following regimen:
  Placebo Patients < 45 kg - 3 tablets 3 times a day with meals
  Placebo Patients > 45 kg - 5 tablets 3 times a day with meals
  Idebenone: All PROTI patients randomised to idebenone treatment will receive high dose idebenone. This is defined according to body weight. In patients weighing 45 kg or less, it is 1350 mg/day (3 x 150 mg tablets three times per day with meals). In patients weighing more than 45 kg, it is 2250 mg/day (5 x 150 mg tablets three times per day with meals).
- Idebenone: Following the body weight, patients will be allocated to one of the following regimen:
  Idebenone Patients < 45 kg - 3 tablets 3 times a day with meals
  Idebenone Patients > 45 kg - 5 tablets 3 times a day with meals
  Idebenone: All PROTI patients randomised to idebenone treatment will receive high dose idebenone. This is defined according to body weight. In patients weighing 45 kg or less, it is 1350 mg/day (3 x 150 mg tablets three times per day with meals). In patients weighing more than 45 kg, it is 2250 mg/day (5 x 150 mg tablets three times per day with meals).
Period: Overall Study
Arm/Group | Placebo | Idebenone
Started | 13 | 16
Completed | 13 | 15
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Idebenone | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (16.5) | 35.8 (16.9) | 37.1 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  Germany | 3 | 5 | 8
  United Kingdom | 7 | 7 | 14
  Austria | 2 | 2 | 4
  Netherlands | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Patient Assessment of Treatment Assignment: Comparison of the Proportions of Patients Randomised to Idebenone and Placebo Who Assessed That They Received Idebenone
Description: The primary efficacy endpoint was the comparison of the number of patients randomized to idebenone and placebo, who assessed that they received idebenone treatment.
Time Frame: At 2 months after study start
Measure: Number; unit: participants
Arm/Group | Placebo | Idebenone
Number analyzed (Participants) | 13 | 16
participants | 6 | 8

2. Secondary Outcome: Comparison of the Percentage of Participants Randomised to Idebenone and Placebo Who Withdrew Early Due to Recurrence or Worsening of FRDA Symptoms
Description: There was no Withdrawal due to recurrence or worsening of FRDA symptoms
Time Frame: Within 2 months (i.e. Early withdrawal visit)
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Idebenone
Number analyzed (Participants) | 13 | 16
percentage of patients | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Idebenone
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/16
Other Adverse Events (participants affected / at risk) | 9/13 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Idebenone (N=16)
Fractured femur (Injury, poisoning and procedural complications) | 0 | 1
Dislocated hip (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Idebenone (N=16)
Fall (Injury, poisoning and procedural complications) | 3 | 3
Fatigue (General disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 2
Speech disorder (Nervous system disorders) | 2 | 2
Pain (General disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Parathyroid gland enlargement (Endocrine disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No